CLINICAL TRIAL: NCT02147444
Title: Multi-center, Prospective, Non-interventional, Observational Cohort Study to Investigate Effectiveness and Safety of Rivaroxaban on Prevention of Stroke and Systemic Embolism in Patients With Non-valvular Atrial Fibrillation in Japanese Clinical Practice
Brief Title: Evaluation of Effectiveness and Safety of Xa Inhibitor for the Prevention of Stroke And Systemic Embolism in a Nationwide Cohort of Japanese Patients Diagnosed as Non-valvular Atrial Fibrillation
Acronym: EXPAND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tohoku University (Other)
Responsible Party: Principal Investigator, Hiroaki Shimokawa, MD, PhD, MD, PhD, Department of Cardiovascular Medicine, Tohoku University
Other Study IDs: EXPAND study; UMIN000009376 (Other: UMIN)
Record Dates: First submitted 2014-05-12; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Rivaroxaban; Non-valvular atrial fibrillation; NOAC; Xa inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-valvular atrial fibrillation: * Patients diagnosed with non-valvular atrial fibrillation
  * Patients who are treated or will be treated with rivaroxaban

SUMMARY:
The efficacy and safety of a novel oral Xa inhibitor for stroke and systemic embolism, namely rivaroxaban, in non-valvular atrial fibrillation patients are evaluated in Japanese clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the criteria below

* Patients aged over 20 years
* Patients diagnosed with non-valvular atrial fibrillation
* Patients who are treated or will be treated with rivaroxaban
* Patients from whom written informed consent has been obtained

Exclusion Criteria:

Patients who meet any of the criteria below

* The following patients in whom rivaroxaban is contraindicated for use
* Patients with a history of allergies to the ingredients contained in this drug
* Patients having a hemorrhagic event (intracranial hemorrhage, gastrointestinal hemorrhage or other clinically significant hemorrhagic events)
* Patients having liver disease complicated with coagulation disorder or those having moderate or worse liver disorder (Grade B or C in accordance with the Child-Pugh classification)
* Patients having renal failure (creatinine clearance: <15 mL/min)
* Women who are or are likely to be pregnant
* Patients who are treated with HIV protease inhibitors (including ritonavir, atazanavir and indinavir)
* Patients who are treated with oral or injectable formulations of azole antifungal drugs (including itraconazole, voriconazole and ketoconazole (excluding fluconazole))

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-valvular atrial fibrillation (In the present study, non-valvular atrial fibrillation refers to atrial fibrillation without a history of prosthetic valve replacement or mitral valve stenosis.)
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Combinations of symptomatic stroke (ischemic or hemorrhagic) and systemic embolism | up to March/2016
  Primary efficacy endpoint
Clinically significant hemorrhagic events (massive hemorrhage in accordance with the ISTH classification) | up to March/2016
  Primary safety endpoint

SECONDARY OUTCOMES:
Combinations of symptomatic stroke (ischemic or hemorrhagic), systemic embolism, myocardial infarction and cardiovascular death | up to March/2016
  Secondary efficacy endpoints
Symptomatic ischemic stroke | up to March/2016
  Secondary efficacy endpoints
Symptomatic hemorrhagic stroke | up to March/2016
  Secondary efficacy endpoints
Systemic embolism | up to March/2016
  Secondary efficacy endpoints
Acute myocardial infarction/unstable angina pectoris | up to March/2016
  Secondary efficacy endpoints
Cardiovascular death | up to March/2016
  Secondary efficacy endpoints
Deep vein thrombosis/pulmonary thromboembolism | up to March/2016
  Secondary efficacy endpoints
Transient ischemic attack | up to March/2016
  Secondary efficacy endpoints
Interventional/surgical treatment | up to March/2016
  Secondary efficacy endpoints
All-cause death | up to March/2016
  Secondary efficacy endpoints
Clinically insignificant hemorrhagic events (hemorrhagic events other than clinically significant hemorrhagic events) | up to March/2016
  Secondary safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Shimokawa, MD, PhD, Study Chair — Department of Cardiovascular Medicine, Tohoku University Graduate School of Medicine
Locations (1):
- Department of Cardiovascular Medicine, Tohoku University Graduate School of Medicine, Sendai, Miyagi, Japan

REFERENCES:
- See also: EXPAND study home page — http://cms.captool.jp/expand/